CLINICAL TRIAL: NCT02247713
Title: An International Study on the Use of PET/CT in Radiotherapy Planning in Low and Middle Income Countries
Acronym: PERTAIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Other Study IDs: M14PRI
Record Dates: First submitted 2014-08-14; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Non Small Cell Lung Cancer Stage III
Keywords: PET; radiotherapy; international; NSCLC; overall survival; low and middle income countries
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective cohort: Participating centers will retrospectively provide demographic, tumor, treatment and follow-up details on at least 25 consecutive patients with stage III NSCLC previously treated with curative intent chemoradiotherapy (concurrent or sequential) in the period between 2010 and 2013.
- Prospective cohort: Participating centers will provide prospective data on patients with stage III NSCLC treated with curative intent concurrent chemoradiotherapy. Centers will be asked to include at least 25 consecutive cases following the training intervention and the successful local implementation of PET/CT for RTP in NSCLC.

SUMMARY:
A part retrospective, part prospective cohort study to assess the difference in 2-year overall survival in patients with stage III NSCLC receiving chemoradiotherapy with curative intent in low and middle income countries before and after a training intervention on the use of PET/CT for radiotherapy treatment planning.

DETAILED DESCRIPTION:
Over the years, the incidence of lung cancer has risen in some low and middle income countries due to the rise in tobacco use. Patients commonly present with lung cancer in an advanced stage (stage III and IV) are not suitable for surgical resection, but may be considered for radiotherapy. For patients in those countries who are not suitable for surgical resection, radiotherapy offers the best chance of cure, best improvement in local cancer control, best palliation and fewest side-effects. For accurate patient selection for curative treatment and accurate staging of lung cancer, the use of fused 18F-fluorodeoxyglucose Positron Emission Tomography/ Computed Tomography (FDG PET/CT) imaging has been shown to be superior to CT alone. It has also been shown to have a significant impact when used in the radiation treatment planning process and in particular for when used for target volume delineation, where a significant reduction in interobserver variation has been noted.

In recent years, many health care institutions in low and middle income countries have established Nuclear Medicine (NM) imaging in routine clinical practice in conjunction with modern Radiation Oncology (RO) facilities. The installation of hybrid PET/CT systems in these countries permits more the increased use of PET/CT for both staging and radiotherapy planning. However the successful implementation of PET/CT for radiotherapy planning (RTP) requires a degree of expertise to safely and accurately implement this imaging technique. A recently published review by the International Atomic Energy Agency (IAEA), about current trends in NM in developing countries showed there is still lack of expertise, equipment and human resources to gain benefit from this imaging technique. In RO, difficulties in the implementation of this technique are mainly related to inadequate training of staff and lack of local expertise.

Quality assurance of the PET/CT scanners might be compromised when not performed according to accepted nuclear medicine quality assurance standards. Therefore, there is a concern that, if used without appropriate training or expertise, suboptimal image quality may result and inappropriate interpretation of the PET/CT for RTP may occur. In this study to help provide PET Quality Control will be executed to aim for a standardized PET image quality that meets the minimum requirements of European Association of Nuclear Medicine standards. Participating centers will be assisted to earn the European Association of Nuclear Medicine (EANM) Research Ltd (EARL) accreditation. The quality of the imaging can be influenced by physiological and technical factors. The Standardized Uptake Value (SUV) allows for semi quantitative evaluation in PET imaging, and is influenced by these factors. Spatial resolution affects SUV values significantly and this parameter can differ a lot between multiple centers. The EANM NEMA NU 2001/2007 2 Image Quality Phantom allows for standardization of PET imaging between centers with different scanners, using the activity coefficient recovery curve (ACRC) as a parameter for quantification of this spatial resolution.

It is already known that FDG PET/CT based RTP enables appropriate selection of patients who will benefit from curative radiation therapy. One possible cause of failure in radiotherapy is the inability to accurately define the tumor edges. In these patients there are no other possible curative salvage treatment options and the disease is incurable. It is hoped that FDG PET/CT based RTP will improve tumor volume delineation (TVD) and hence improve outcomes following curative radiotherapy. There is also clear evidence that PET/CT standardizes TVD in patients with NSCLC. However, what is not known is the impact of PET/CT based TVD on patient outcomes such as survival as distinct from the benefit of PET/CT for patient selection for curative treatment. Furthermore, the impact of a training intervention on the use of PET/CT RTP in 2-year overall survival has not been studied to the best of our knowledge.

This study will evaluate the possible impact of the use of PET/CT for TVD on 2-year overall survival in patients with stage III NSCLC referred for curative intent radiotherapy with chemotherapy in low and middle income countries, this study involves a retrospective cohort study, a training intervention, and a prospective cohort study. The training intervention will focus on standard FDG PET/CT acquisition, FDG PET/CT image quality, staging procedure for FDG PET/CT acquisition and FDG PET/CT for RTP acquisition and Tumor Volume Delineation.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed NSCLC
* stage III as per local diagnostic protocol or agreement of local multidisciplinary team
* available for clinical follow-up for at least 2 years
* suitable for treatment with a radical target volume in the opinion of a radiation oncologist
* ECOG performance 0 or 1
* signed informed consent
* ability to commence radiation therapy within 4 weeks of acquisition of the RTP PET/CT
* suitable for concurrent chemoradiotherapy (prospective cohort only)

Exclusion Criteria:

* other neoplasms in the last 5 years except non-melanoma skin cancer
* stage IV disease diagnosed before acquisition of staging PET/CT
* inability to provide informed consent
* uncontrolled diabetes mellitus
* pregnant or breast feeding mothers
* tuberculosis
* neo-adjuvant chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The retrospective cohort study includes at least 250 patientswith stage III NSCLC with curative intent chemoradiotherapy (sequential or concurrent), 125 patients in the first arm (non PET staged) and 125 patients (PET staged) in the second arm. The prospective cohort study includes at least 250 patients (PET staged) receiving concurrent chemoradiotherapy based on PET/CT RTP. In total, we aim to include a number of 519 patients.
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival | the included patients will be followed for a maximum of 2 years
  Determine the impact of PET/CT in RTP on 2-year overall survival rates for patients with stage III NSCLC receiving chemoradiotherapy with curative intent. Patients from the retrospective cohort will be selected from the institutional database and were treated between 2010 to 2013. Patients from the prospective cohort will be selected until the end of 2015.

SECONDARY OUTCOMES:
Observer agreement with expert contours as a measure of the effect of a training intervention on tumor volume delineation | up to 5 months
  Determine the impact of a PET/CT in RTP training intervention on tumor volume delineation for stage III NSCLC radiotherapy. Different parameters are used to determine the observer variation: Dice Index, median surface distances
Baseline PET/CT characteristics as a measure for PET/CT scanner performance | up to 8 months
  Determine the quality of PET/CT scanners. Study baseline PET/CT imaging protocols and image acquisition characteristics with the following parameters: recovery coefficients, spatial resolution measurement, and calibration of SUV determination. All centers will participate in the EARL accreditation programme.

CONTACTS AND LOCATIONS:
Overall Officials: Wouter V Vogel, MD, Principal Investigator — Antoni van Leeuwenhoek - Netherlands Cancer Institute; Gerard G Hanna, MD, Principal Investigator — Centre for Cancer Research and Cell Biology, Queen's University Belfast